CLINICAL TRIAL: NCT01662089
Title: A Pilot Study of the Efficacy in Treatment of Female Pattern Hair Loss Using 5% Minoxidil Solution Combinded With Oral Chelated Zinc Supplement
Brief Title: The Efficacy in Treatment of Female Pattern Hair Loss Using 5% Minoxidil Solution Combinded With Zinc Supplement
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Associate Professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SirirajH-004
Record Dates: First submitted 2012-08-05; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Female Pattern Alopecia
Keywords: Female pattern hair loss
MeSH Terms: conditions — Alopecia | interventions — Zinc; Starch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chelate zinc suppliment (Experimental): 15mg Chelate zinc suppliment : additional to standard 5% minoxidil
  Interventions: Drug: 15 mg Chelate zinc supplement
- Placebo drug (Placebo Comparator): Placebo drug to compare with 15mg chelated Zn : additional to standard 5% minoxidil
  Interventions: Drug: Placebo drug supplement

INTERVENTIONS:
Drug: 15 mg Chelate zinc supplement — 15 mg Chelate zinc additional to standard 5% minoxidil
  Other Names: zinc, Zn
  Arms: Chelate zinc suppliment
Drug: Placebo drug supplement — Placebo drug instead of Zinc supplement
  Other Names: starch
  Arms: Placebo drug

SUMMARY:
Zinc supplement is a popular trace element gave to Female pattern hair loss (FPHL) patient. But the type of patient, efficacy, and side effect in detail of zinc supplement are not well characterized. The purpose of this study is to determine efficacy and side effect of chelated zinc in FPHL who using 5%minoxidil solution.

DETAILED DESCRIPTION:
5%minoxidil solution is standard treatment for Female pattern hair loss (FPHL) patient. We gave 15mg chelate Zinc / Placebo drug to patient as an additional trace element. Then measure growth of hair by Global photograph, Microscope hair count, micrometer and record case and side effect during 10 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female Pattern Hair Loss ( Ludwig classification grade 1 and 2 )

Exclusion Criteria:

* Underlying disease ; Anemia, Diabetes, chronic alcoholism, previous gastrointestinal surgery, short bowel syndrome, Crohn's disease, digestive disorder, hypo/hyperthyroidism, sickle cell disease, autoimmune disease, iron deficiency
* Psychologic disorder trichotillomania
* Diet control
* Pregnancy or lactation
* On supplement diet within 3 month prior to trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Compare clinical improvement before and after treatment | 6 month
  Measure clinical by Global photographic view using 7 point scale. Review picture by 2 dermatologist
Compare hair density before and after treatmen | 6 month
  Measure Hair density by microscope photo of area 1 cm2. Conut number of hair in photo.
Compare average hair shaft diameter before and after treatment | 6 month
  Compare average hair shaft diameter before and after treatment Measure hair shaft diameter using electronic outside micrometer.

SECONDARY OUTCOMES:
Number of pateint with Side effect | 6 month
  Using side effect record form to record side effect from treatment Count number of pateint with side effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok, Thailand